CLINICAL TRIAL: NCT01231828
Title: Method of Assessment of Driving Ability in Patients Suffering From Wakefulness Pathologies. Impact of Lactulose and Carnitine Treatment.
Brief Title: Method of Assessment of Driving Ability in Patients Suffering From Wakefulness Pathologies.
Acronym: AutoSop-Foie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A90591-34
Record Dates: First submitted 2010-10-04; First posted 2010-11-01 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Cirrhosis
Keywords: sleep; cirrhosis; encephalopathy; simulated driving; sleep disorders
MeSH Terms: conditions — Fibrosis; Brain Diseases; Sleep Wake Disorders | interventions — Carnitine; Lactulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carnitine (Experimental): Versus placebo.
  Interventions: Drug: L-carnitine
- Lactulose (Experimental): Versus placebo
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: L-carnitine — L-carnitine 4g per day (4 bottles of 10ml).
  Other Names: Levocarnil.
  Arms: Carnitine
Drug: Lactulose — Lactulose (30-60 ml per day)
  Other Names: Duphalac.
  Arms: Lactulose

SUMMARY:
The project will improve scientific knowledge regarding a recent law applying potentially to every french driver. It will give for the first time an indication on the impact of alerting treatments on driving risks. It will reinforce the links between different research environments (sleep physiopathology, clinical research, cognitive neurosciences, drivers supervision, virtual reality, pharmacology) among the "Réseau Eveil Sommeil Attention et Transports" (RESAT) network.

DETAILED DESCRIPTION:
Excessive daytime sleepiness is responsible of 20% of traffic accidents and 2/3 of truck accidents on French Freeways. Since the publication of a new law (2005 december 28th - Official Journal) regulating fitness to drive, the Maintenance of Wakefulness Test (MWT) is now mandatory to evaluate driving skills of patients suffering of excessive daytime sleepiness. The MWT has shown a good predictability of driving handicap on simulators in patients suffering from obstructive sleep apnea syndrome. Nevertheless no study has proven yet the predictability of the MWT regarding real and simulated driving in patients suffering from hepatic encephalopathy. Furthermore, even if therapeutic drugs significantly improve MWT scores there is no data available concerning the impact of these drugs on fitness to drive. Lactulose, a treatment of hepatic encephalopathy, has not been tested as a counter measure to driving impairment. This lack of knowledge is a major handicap to evaluate driving skills of treated patients suffering from excessive daytime sleepiness. The main objective of our project is to test the predictive value of the MWT on real and simulated driving performances in untreated and treated sleepy patients suffering from hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis proved by histologic or clinico-biologics criteria, whatever its severity, its stability defined by a child stable score (variation < 2 points for the last month) without any other disease which could be responsible of excessive daytime sleepiness
* driver's licence since at least 2 years
* driving more than 2000 Km/year
* registered to French national health and pensions organization
* having given their written light agreement in order to participate in the study.

Exclusion Criteria:

* Night workers
* neurologic disease
* recent strong complication (< 30 days)
* recent antibiotics or lactulose intake
* substance abusers (alcohol)
* hepatoma more than 5 cm
* disorder associated which engaged life prognostic in a short time
* glycemia fasted > 8 mmol/l
* haemoglobin < 10g/l
* neurologic or psychiatric disorders associated which affect superiors functions,
* hepatic encephalopathy stage 3 or 4
* having participated in a clinical study during the last 6 months
* drugs abusers
* unable to drive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sleep latency during Maintenance of Wakefulness Test (MWT) | 40 min

SECONDARY OUTCOMES:
Nocturnal sleep quality and quantity will be measured by Polysomnography (PSG). | 1 night
Nocturnal sleep quality and quantity measured by Actimetry. | during 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Astrid PIQUET, Principal Investigator — University Hospital, Caen; Thong DAO, Study Director — University Hospital, Caen
Locations (1):
- University Hospital of Caen, Caen, France